CLINICAL TRIAL: NCT00949286
Title: Action in Diabetes and Vascular Disease Preterax and Diamicron MR Controlled Evaluation Post Trial Observational Study
Acronym: ADVANCE-ON
Status: Completed | Type: Observational
Sponsor: The George Institute (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Other Study IDs: ADVANCE-ON
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to determine the long term, post trial effects of the two interventions studied in ADVANCE (routine blood pressure lowering with perindopril-indapamide as compared with placebo and intensive gliclazide-MR based glucose control as compared to standard guideline based glucose control) in individuals with type 2 diabetes at high risk of cardiovascular events. The long term, post randomization effects of the two study interventions will be investigated separately as they were for the main trial. This study will clarify and quantify the long-term, post trial (often referred to as legacy) effects of these two interventions in a broader population of patients with type 2 diabetes from high and low to middle income countries, and in the setting of comprehensive cardiovascular risk factor treatment. With the ADVANCE trial infrastructure and surveillance system already in place, the implementation of extended follow-up will be feasible. The conclusions of this follow up study will have profound clinical implications for the care of patients with type 2 diabetes around the world.

DETAILED DESCRIPTION:
The long term, post randomization effects of the two study interventions will be investigated separately as they were for the main trial. This study will clarify and quantify the long-term, post trial (often referred to as legacy) effects of these two interventions in a broader population of patients with type 2 diabetes from high and low to middle income countries, and in the setting of comprehensive cardiovascular risk factor treatment. With the ADVANCE trial infrastructure and surveillance system already in place, the implementation of extended follow-up will be feasible. The conclusions of this follow up study will have profound clinical implications for the care of patients with type 2 diabetes around the world.

ELIGIBILITY:
Inclusion Criteria:

* Participated in ADVANCE
* Ability to provide informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All living participants who took part in the ADVANCE study
Sampling Method: Non-Probability Sample
Enrollment: 8494 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Major macrovascular events -a composite of non-fatal myocardial infarction, non-fatal stroke and death from any cardiovascular cause (based on investigator diagnosis) | 2014
Death from any cause | 2014

SECONDARY OUTCOMES:
Death from any cardiovascular cause | 2014
Major clinical microvascular events - a composite of requirement for renal replacement therapy, death from renal disease and development of severe diabetes-related eye disease | 2014
Composite of major macrovascular events and major clinical microvascular events | 2014
Stroke (non-fatal and fatal) | 2014
Requirement for renal replacement therapy (dialysis or transplantation) | 2014
Death from renal disease | 2014
Development of severe diabetes-related eye disease defined as the requirement for retinal photocoagulation or similar treatment and development of diabetes-related blindness in either eye in a participant known not to have this condition at study entry | 2014
Major hypoglycaemia - an episode associated with transient central nervous system dysfunction without other apparent cause in which the individual was unable to treat him/herself and had help from another person to administer glucose or glucagon | 2014
Myocardial infarction (non-fatal and fatal) | 2014

CONTACTS AND LOCATIONS:
Overall Officials: John P Chalmers, Principal Investigator — The George Institute; Stephen MacMahon, Principal Investigator — The George Institute
Locations (172):
- Australia (22):
  - LCC 80 - Canberra Hospital, Garran, Australian Capital Territory
  - LCC 28 - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - LCC 48 - Gosford, Gosford, New South Wales
  - LCC 59 - Liverpool Hospital, Liverpool, New South Wales
  - LCC 78 - Wentworth Diabetes Centre, Penrith, New South Wales
  - LCC 56 - Prince of Wales Hospital, Randwick, New South Wales
  - LCC 55 - Royal North Shore Hospital, St Leonards, New South Wales
  - LCC 23 - Wollongong Hospital, Wollongong, New South Wales
  - LCC 24 - Mater Hospital, Brisbane, Queensland
  - LCC 42 - Princess Alexandra Hospital, Brisbane, Queensland
  - LCC 74 - Redcliffe Hospital, Redcliffe, Queensland
  - LCC 43 - Gold Coast Hospital, Southport, Queensland
  - LCC 114 - Townsville Mater Hospital, Townsville, Queensland
  - LCC 73 - Repatriation General Hospital, Daw Park, South Australia
  - LCC 66 - Lyell McEwin Health, Elizabeth Vale, South Australia
  - LCC 61 - Launceston General Hospital, Launceston, Tasmania
  - LCC 65 - Dandenong Hospital, Dandenong, Victoria
  - LCC 33 - The Northern Hospital, Epping, Victoria
  - LCC 32 - Austin & Repatriation Hospital, Heidelburg, Victoria
  - LCC 76 - The Alfred Hospital, Melbourne, Victoria
  - LCC 109 - Rural Clinical Trials Research Unit, Shepparton, Victoria
  - LCC 50 - Fremantle Hospital, Fremantle, Western Australia
- Canada (10):
  - LCC 468 - Calgary Metabolic Education and Research Centre, Calgary, Alberta
  - LCC 454 University of British Columbia, Vancouver, British Columbia
  - LCC 467 - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - LCC 465 - St. Joseph's Health Centre, London, Ontario
  - LCC 459 - University of Toronto, Toronto, Ontario
  - LCC 452 - Centre de recherche clinique de Laval, Laval, Quebec
  - LCC 453 - Centre hospitalier de l'Universite de Montreal, Montreal, Quebec
  - LCC 460 - Centre Hospitalier de L'universitaire de Sherbrooke, Sherbrooke, Quebec
  - LCC 466 - Centre de recherche d'endocrinologie, Sherbrooke, Quebec
  - LCC 470 - Hôpital Laval, Ste-Foy, Quebec
- China (49):
  - LCC 643 - 2nd Aff Hospital of Baotou Medical College, Baotou
  - LCC 644 - Baotou Iron & Steel Corporation's Hospital,, Baotou
  - LCC 600 - Center Hospital of Aviation, Beijing
  - LCC 601 - 305 Hospital of Chinese PLA, Beijing
  - LCC 602 - Chinese PLA General Hospital, Beijing
  - LCC 623 - Beijing 306 Hospital, Beijing
  - LCC 626 - First Hospital of Peking University, Beijing
  - LCC 627 - Peking Union Medical College Hospital, Beijing
  - LCC 628 - Capital Steel Hospital, Beijing
  - LCC 629 - Aff Beijing Tongren Hospital, Beijing
  - LCC 630 - Beijing Hypertension League Institute, Beijing
  - LCC 631 - Beijing Jiuxianqiao Hospital, Beijing
  - LCC 632 - Dept Endocrinology Beijing 306 Hospital, Beijing
  - LCC 633 - Cardiovascular Institute & Fu Wai Hospital, Beijing
  - LCC 634 - Beijing Anzhen Hospital, Beijing
  - LCC 637 - Chinese Air Force General Hospital, Beijing
  - LCC 661 - Institute of Gerontology of Benxi City, Benxi
  - LCC 607 - People's Hospital of Binzhou City, Binzhou
  - LCC 609 - Xiang-ya Hospital,, Changsha
  - LCC 620 - Municipal Hospital of Chengdou, Chengdu
  - LCC 657 - The 1st Aff Hospital, Chengdu
  - LCC 610 - Second Affiliated Hospital of Dalian Medical University, Dalian
  - LCC 624 - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - LCC 658 - The 1st Aff Hospital of Guiyang Medical College, Guiyang
  - LCC 641 - The 2nd Aff Hospital of Harbin Medical University, Harbin
  - LCC 653 - Aff Hospital of Anhui Medical University, Hefei
  - LCC 642 - The Institute of Aged Gerontology of Inner Mongolia, Hohhot
  - LCC 606 - Shandong Academy of Medical Sciences,, Jin’an
  - LCC 660 - Shandong Academy of Medical Sciences, Jin’an
  - LCC 622 - The First People's Hospital of Lianyungang City, Lianyungang
  - LCC 654 - The 3rd Aff Hospital of Jiangxi Medical University, Nanchang
  - LCC 655 - The 1st Aff Hospital of Jiangxi Medical College, Nanchang
  - LCC 651 - Jiangsu Institute of Geriatrics,, Nanjing
  - LCC 608 - Qingdao City Hospital, Qingdao
  - LCC 603 - Rujin Hospital, Shanghai
  - LCC 635 -Aff Ruijin Hospital of Shanghai Second Medical University, Shanghai
  - LCC 636 - Chang Zheng Hospital of Shanghai, Shanghai
  - LCC 638 - Shanghai 6th People's Hospital, Shanghai
  - LCC 611 - Hua Tai Hospital, Shenyang
  - LCC 618 - Hebei Academy of Medical Sciences, Shijiazhuang
  - LCC 646 - The 2nd Aff Hospital of Hebei Medical University, Shijiazhuang
  - LCC 613 - Cardiovascular Institute of Shanxi Province, Taiyuan
  - LCC 645 - Hospital of Kailuan, Tangshan
  - LCC 639 - Metabolic Disease Hospital of Tianjin Medical University, Tianjin
  - LCC 640 - 3rd Hospital of Tianjin City, Tianjin
  - LCC 619 - The First Hospital of Ning Bo City Municipal, Xinning
  - LCC 647 - First Hospital of Yang Quan City, Yangquan
  - LCC 614 -The First Affiliated Hospital of Henan Medical University, Zhengzhou
  - LCC 616 - Center Hospital of Zhumadian City, Zhumadian
- Czechia (5):
  - LCC 437 - Metabolicke Centrum, Neratovice
  - LCC 372- Fakultni Nemocnice, Ostrava-Poruba
  - LCC 438 - Diabetologicka ambulance, Písek
  - Lcc 435 - Ikem, Prague
  - LCC 369- Masarykova Nemocnice, Ústí nad Labem
- Estonia (2):
  - LCC 280 - Tallinn Central, Tallinn
  - LCC 281 - Dept of Medicine, Tartu
- France (9):
  - LCC 320 - CHU Angers, Angers
  - LCC 376 - CH Avignon - Hôpital Henri Duffaut, Avignon
  - LCC 375 - CH Nevers, Nevers
  - LCC 373 - CHU Hopital Caremeau, Nîmes
  - LCC 329 - CHU Bichat, Paris
  - LCC 315 - Hôpital Jean Bernard la Miletrie, Poitiers
  - LCC 310 - Hôpital Sud, Rennes
  - LCC 304 - CHU Hôpital Civil, Strasbourg
  - LCC 374 - CHU Hôpital Jeanne d' Arc, Toul
- Germany (2):
  - LCC 377 - Zentrum fur Klinische Studien, Dresden
  - LCC 330 - Klinikyum der Universitat Munchen, Munich
- Hungary (2):
  - LCC 336 - Heart Center Foundation-DRC Ltd, Balatonfüred
  - LCC 335 - Bajcsy Zsilinszky Kórház, Budapest
- India (3):
  - Lcc 740 - Aiims, Delhi
  - LCC 744 - Care Hospital, Hyderabad
  - LCC 741 - Madras Diabetic Research Foundation, Madras
- Ireland (5):
  - LCC 832 - Portincula Hospital, Ballinasloe
  - LCC 514 - Beaumont Hospital, Dublin
  - LCC 810 - Mater Hospital, Dublin
  - LCC 817 - St James Hospital, Dublin
  - LCC 806 - Adelaide & Meadth Hospital, Tallaght
- LCC 418 - Ospedale San Gerado, Milan, Italy
- Lithuania (2):
  - LCC 270 - Institute of Cardiology, Kaunas
  - LCC 273 - Institute Psychophysiology and Rehabilitation, Palanga
- Malaysia (5):
  - LCC 901 - Penang Medical College, George Town
  - LCC 903 - Hospital Ipoh, Ipoh
  - LCC 904 - Universiti Sains Malaysia, Kota Bharu
  - LCC 902 - University of Malaya Medical Centre, Kuala Lumpur
  - Universiti Kebangsaan Malaysia & Universiti Teknologi MARA, Putrajaya
- Netherlands (8):
  - LCC 352 - Justus Medical Research, Eindhoven
  - LCC 354 - Stichting Huisartsen Laboratorium, Etten-Leur
  - LCC 347 - Martini Ziekenhuis, Groningen
  - LCC 850 - Andromed Groningen, Groningen
  - LCC 351 - Andromed Rotterdam, Rotterdam
  - LCC 852 - Andromed Baarn, Rotterdam
  - LCC 851 - Andromed Oost, Velp
  - LCC 356 - Huisartsenpraktijk Tollenslaan, Zeist
- New Zealand (8):
  - LCC 11 - Middlemore Hospital, Auckland
  - LCC 14 - North Shore Hospital, Auckland
  - LCC 12 - Christchurch Hospital, Christchurch
  - LCC 5 - Hawkes Bay Hospital, Hastings
  - LCC 2 - Palmerston North Hospital, Palmerston North
  - LCC 91 - Timaru Hospital, Timaru
  - LCC 6 Waikato Hospital, Waikato
  - LCC 1 - Wellington Hospital, Wellington
- Philippines (4):
  - LCC 909 - Makati Medical Center, Makati City, Manila
  - LCC 906 - Philippine General Hospital, Manila
  - LCC 907 - East Avenue Medical Centre, Quezon City
  - LCC 908 - Diabetes Foundation, Quezon City
- Poland (10):
  - LCC 426 - NZOZ Specjalistyczna Poradnia Endokrynologii, Elblag
  - LCC 382 - Puls Med, Katowice
  - LCC 381 - I Klinika Kardiologii, Krakow
  - LCC 383 - Klinika Chorob Metabolicznych, Krakow
  - LCC 389 - Zakład Angiologii, Krakow
  - LCC 390 - Klinika Choroby Wiencowej, Krakow
  - LCC 380 - I Oddzial Chorob Wewnetrznych, Kutno
  - LCC 392 - Osrodek Diabetologii, Olsztyn
  - LCC 378 - Klinika Nefrologii, Poznan
  - LCC 394 - II Oddzial Chorob Wewnetrznvch, Radom
- Russia (3):
  - LCC 420 - Russian Peoples Friendship University, Moscow
  - LCC 421 - St Petersburg State Medical University, Saint Petersburg
  - LCC 424 - Research Institute of Cardiology, Saint Petersburg
- Slovakia (3):
  - LCC 254 - Poliklinikou Vychod, Košice
  - LCC 252 - Nemocnica s poliklinikou, Levice
  - LCC 253 - Nemocnica s poliklinikou, Lučenec
- United Kingdom (19):
  - LCC 517 - Aberdeen Royal Infirmary, Aberdeen
  - LCC 813 - Monklands Hospital, Airdrie
  - LCC 819 - Royal United Hospital, Bath
  - LCC 815 - City Hospital, Birmingham
  - LCC 821 - West Byfleet Health Centre, Byfleet
  - LCC 594 - Glasgow Royal Infirmary, Glasgow
  - LCC 826 - St Mary's Hospital, Isle of Wight
  - LCC 533 - Leicester Royal Infirmary, Leicester
  - LCC 809 - Royal Liverpool University Hospital, Liverpool
  - LCC 543 - St Mary's, London
  - LCC 511 - Manchester Royal Infirmary, Manchester
  - LCC 829 - Northampton General Hospital, Northampton
  - LCC 830 - George Eliot Hospital, Nuneaton
  - LCC 812 - Royal Alexandra Hospital, Paisley
  - LCC 816 - Peninsula Medical School Headquarters, Plymouth
  - LCC 820 - The Diabetes Centre, Reading
  - LCC 827 - Northern General Hospital, Sheffield
  - Sheffield Hallamshire, Sheffield
  - LCC 831 - Warwick General Hospital, Warwick

REFERENCES:
- [Background] Patel A; ADVANCE Collaborative Group; MacMahon S, Chalmers J, Neal B, Woodward M, Billot L, Harrap S, Poulter N, Marre M, Cooper M, Glasziou P, Grobbee DE, Hamet P, Heller S, Liu LS, Mancia G, Mogensen CE, Pan CY, Rodgers A, Williams B. Effects of a fixed combination of perindopril and indapamide on macrovascular and microvascular outcomes in patients with type 2 diabetes mellitus (the ADVANCE trial): a randomised controlled trial. Lancet. 2007 Sep 8;370(9590):829-40. doi: 10.1016/S0140-6736(07)61303-8. PMID 17765963
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Derived] Wang N, Harris K, Hamet P, Harrap S, Mancia G, Poulter N, Williams B, Zoungas S, Woodward M, Chalmers J, Rodgers A. Cumulative Systolic Blood Pressure Load and Cardiovascular Risk in Patients With Diabetes. J Am Coll Cardiol. 2022 Sep 20;80(12):1147-1155. doi: 10.1016/j.jacc.2022.06.039. PMID 36109108
- [Derived] Oshima M, Jun M, Ohkuma T, Toyama T, Wada T, Cooper ME, Hadjadj S, Hamet P, Harrap S, Mancia G, Marre M, Williams B, Chalmers J, Woodward M, Perkovic V; ADVANCE Collaborative Group. The relationship between eGFR slope and subsequent risk of vascular outcomes and all-cause mortality in type 2 diabetes: the ADVANCE-ON study. Diabetologia. 2019 Nov;62(11):1988-1997. doi: 10.1007/s00125-019-4948-4. Epub 2019 Jul 13. PMID 31302707
- [Derived] Mohammedi K, Woodward M, Hirakawa Y, Zoungas S, Colagiuri S, Hamet P, Harrap S, Poulter N, Matthews DR, Marre M, Chalmers J; ADVANCE Collaborative Group. Presentations of major peripheral arterial disease and risk of major outcomes in patients with type 2 diabetes: results from the ADVANCE-ON study. Cardiovasc Diabetol. 2016 Sep 2;15(1):129. doi: 10.1186/s12933-016-0446-x. PMID 27590190
- [Derived] Wong MG, Perkovic V, Chalmers J, Woodward M, Li Q, Cooper ME, Hamet P, Harrap S, Heller S, MacMahon S, Mancia G, Marre M, Matthews D, Neal B, Poulter N, Rodgers A, Williams B, Zoungas S; ADVANCE-ON Collaborative Group. Long-term Benefits of Intensive Glucose Control for Preventing End-Stage Kidney Disease: ADVANCE-ON. Diabetes Care. 2016 May;39(5):694-700. doi: 10.2337/dc15-2322. Epub 2016 Mar 22. PMID 27006512
- [Derived] Zoungas S, Chalmers J, Neal B, Billot L, Li Q, Hirakawa Y, Arima H, Monaghan H, Joshi R, Colagiuri S, Cooper ME, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Lisheng L, Mancia G, Marre M, Matthews DR, Mogensen CE, Perkovic V, Poulter N, Rodgers A, Williams B, MacMahon S, Patel A, Woodward M; ADVANCE-ON Collaborative Group. Follow-up of blood-pressure lowering and glucose control in type 2 diabetes. N Engl J Med. 2014 Oct 9;371(15):1392-406. doi: 10.1056/NEJMoa1407963. Epub 2014 Sep 19. PMID 25234206